CLINICAL TRIAL: NCT01593033
Title: Randomized, Double-blind, Placebo-controlled Trial Evaluating the Impact of Micronutrient Supplementation and Fish Oil + Micronutrient Supplementation in the Treatment of Sub-clinical Environmental Enteropathy in Rural Malawian Children
Brief Title: Effectiveness of Micronutrient Supplementation and Fish Oil + Micronutrient Supplementation in the Treatment of Environmental Enteropathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MJM - Fish Oil
Record Dates: First submitted 2012-05-03; First posted 2012-05-07 (Estimated); Last update posted 2013-01-14 (Estimated); Status verified 2013-01

CONDITIONS: Environmental Enteropathy
MeSH Terms: interventions — Fish Oils

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (3):
- Fish oil and Micronutrient Supplementation (Experimental)
  Interventions: Dietary Supplement: Fish oil and Micronutrient Supplementation
- Micronutrient Supplementation (Experimental)
  Interventions: Dietary Supplement: Micronutrient Supplement
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Dietary Supplement: Fish oil and Micronutrient Supplementation — 0.9 mL highly purified fish oil (200 mg docosahexaenoic acid, 300 mg eicosapentaenoic acid) to be given daily for 6 months
  1 RDA of all known micronutrients needed for normal child growth in powder form to be given daily for 6 months
  Arms: Fish oil and Micronutrient Supplementation
Dietary Supplement: Micronutrient Supplement — 1 RDA all known micronutrients needed for normal child growth to be given daily in powder form for 6 months 0.9 mL palm oil given daily for 6 months
  Arms: Micronutrient Supplementation
Drug: Placebo — 10 g sugar in granule form to be given daily for 6 months 0.9 mL palm oil to be given daily for 6 months
  Arms: Placebo

SUMMARY:
The purpose of this study is to investigate the therapeutic effectiveness of micronutrients (full RDA) and micronutrients + fish oil as separate interventions in restoring normal gut absorptive and immunological function as measured by the dual sugar permeability test and additional biomarkers in 1-3 year old rural Malawian children at high risk for Environmental Enteropathy.

ELIGIBILITY:
Inclusion Criteria:

* 1-3 years of age
* Lives in study villages
* Will not move in next 6 months
* Caregiver willing to give intervention daily for 6 months

Exclusion Criteria:

* Unable to drink 20 mL of sugar water
* Demonstrating evidence of severe acute malnutrition, WHZ < or = -3, presence of bi-pedal pitting edema
* Apparent need for acute medical treatment for an illness or injury
* Caregiver refusal to participate and return for 3 and 6 month follow-ups

Ages: 1 Year to 3 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 225 (Actual)
Dates: Start 2012-05; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Changes in urine lactulose:mannitol (L:M) ratio following therapy course. | 3 months, 6 months

SECONDARY OUTCOMES:
Changes in the expression of several fecal mRNAs | 3 months, 6 months
Changes in amounts of lactulose and mannitol excreted in the urine as a percentage of the amounts ingested | 3 months, 6 months
Change in height | 3 month, 6 month

CONTACTS AND LOCATIONS:
Overall Officials: Mark J Manary, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Saint Louis Nutrition Project, Blantyre, Malawi

REFERENCES:
- [Derived] Smith HE, Ryan KN, Stephenson KB, Westcott C, Thakwalakwa C, Maleta K, Cheng JY, Brenna JT, Shulman RJ, Trehan I, Manary MJ. Multiple micronutrient supplementation transiently ameliorates environmental enteropathy in Malawian children aged 12-35 months in a randomized controlled clinical trial. J Nutr. 2014 Dec;144(12):2059-65. doi: 10.3945/jn.114.201673. Epub 2014 Oct 1. PMID 25411039